CLINICAL TRIAL: NCT04162093
Title: Preliminary Report Following A Modified Uretero-Ileal Anastomosis in An Ileal Neobladder Combining Wallace Technique With an Extramural Subserous Tunnel in a Single Trough: Our Initial Short-term Results
Brief Title: New Technique for Uretero-ileal Anastomosis for Patient With Bladder Cancer Who Are Suitable for Orthotopic Neobladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hossam Elawady, lecturer of urology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: new uretero-ileal anastomosis
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Orthotopic diversion; Wallace; sub-serous extramural tunnel.
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: the new technique was observed in a group of patients for effectiveness and complications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single trough (Experimental)
  Interventions: Procedure: uretero ileal anastomosis in single trough

INTERVENTIONS:
Procedure: uretero ileal anastomosis in single trough
  Other Names: combining wallace and subserous tunnel in uretero ileal anastomosis

SUMMARY:
there are many techniques for uretero-ileal anastomosis some of them are antirefluxing for protection of the upper urinary tract with many complications including strictures and pyelonephritis with difficult technical issues and long operation time so a modified technique combining the 2 ureter by wallace technique and implanted them in a single trough in the neobladder making the surgery easier and shorter.

this technique was done after informed consent in 45 patients with muscle invasive bladder cancer candidate for radical cystectomy and ileal neobladder diversion

DETAILED DESCRIPTION:
This was a prospective study conducted from 2014 to 2017 in Ain shams university, 73 patients were enrolled from outpatient clinic diagnosed with muscle invasive bladder cancer and candidate for radical cystectomy and orthotopic urinary diversion, 45 patients were included according to patient's acceptance and the inclusion and exclusion criteria.

After having a written informed consent, all selected patients were assessed by detailed history and physical examination, contrast enhanced pelvi-abdominal Computed tomography (CT) scan (for patients with serum creatinine <1.5 mg/dl). Laboratory investigations in the form of complete blood count, coagulation profile, electrolytes, renal and liver function tests. Bowel preparation was done to all patients one or two days before operation.

Cases were diverted using a U-shaped pouch with uretero-ileal anastomosis done in a single trough combining the extramural serous-lined tunnel and Wallace techniques.

ELIGIBILITY:
The inclusion criteria:

* Patients with invasive bladder cancer (T2, T3).
* good performance status
* patients with serum creatinine ≤ 2 mg/dL
* prostatic urethra free of tumor.
* willing to adhere to the follow up regimen.

The exclusion criteria:

* patients not fit for surgical intervention.
* patients with renal or hepatic dysfunction.
* male patients with positive urethral biopsy or diffuse CIS.
* female patients with bladder neck or vaginal involvement.
* concomitant pathological condition in the distal ureters necessitating the excision of a significant segment that hinders proper fashioning of uretero-ileal anastomosis.
* Cases with markedly dilated ureters.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
the rate of vesicoureteral reflux (VUR) | after 6 months and after one year
  the incidence of occurrence of reflux in the patients was assessed
the incidence of anastomotic stricture | after 6 months and after one year
  the incidence of occurrence of uretero ileal stricture in the patients was recorded
the post operative changes in the mean serum creatinine level | after 6 months and after one year
  the change in mean serum creatinine level of the patients was assessed

SECONDARY OUTCOMES:
the incidence of pyelonephritis | after 6 months and after one year
the incidence of urinary incontinence | after 6 months and after one year
the mean operative time of urinary diversion | at the time of the operation
  the time elapsing from bowel selection till the beginning of wound closure

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: after publication
Access Criteria: by the mail of central contact person

REFERENCES:
- [Background] Elawady H, Mahmoud MA, Mostafa DM, Abdelmaksoud A, Safa MW, Elia RZ. Computed tomography virtual cystoscopy for follow-up of patients with superficial bladder tumours in comparison to conventional cystoscopy: An exploratory study. Arab J Urol. 2016 Jul 25;14(3):192-7. doi: 10.1016/j.aju.2016.06.003. eCollection 2016 Sep. PMID 27547459
- [Background] Fakhr I, Mohamed AM, Moustafa A, Al-Sherbiny M, Salama M. Neobladder long term follow-up. J Egypt Natl Canc Inst. 2013 Mar;25(1):43-9. doi: 10.1016/j.jnci.2013.01.001. Epub 2013 Feb 9. PMID 23499206
- [Background] Taub DA, Dunn RL, Miller DC, Wei JT, Hollenbeck BK. Discharge practice patterns following cystectomy for bladder cancer: evidence for the shifting of the burden of care. J Urol. 2006 Dec;176(6 Pt 1):2612-7; discussion 2617-8. doi: 10.1016/j.juro.2006.07.150. PMID 17085172
- [Background] Shigemura K, Yamanaka N, Imanishi O, Yamashita M. Wallace direct versus anti-reflux Le Duc ureteroileal anastomosis: comparative analysis in modified Studer orthotopic neobladder reconstruction. Int J Urol. 2012 Jan;19(1):49-53. doi: 10.1111/j.1442-2042.2011.02870.x. Epub 2011 Oct 17. PMID 22004164
- [Background] Chang DT, Lawrentschuk N. Orthotopic neobladder reconstruction. Urol Ann. 2015 Jan-Mar;7(1):1-7. doi: 10.4103/0974-7796.148553. PMID 25657535
- [Background] Hassan AA, Elgamal SA, Sabaa MA, Salem KA, Elmateet MS. Evaluation of direct versus non-refluxing technique and functional results in orthotopic Y-ileal neobladder after 12 years of follow up. Int J Urol. 2007 Apr;14(4):300-4. doi: 10.1111/j.1442-2042.2006.01716.x. PMID 17470158
- [Background] Elfayoumy H, Abou-Elela A, Orban T, Emran A, Elghoneimy M, Morsy A. A novel antireflux technique for orthotopic ileal bladder substitutes-flat-segment technique: preliminary results. ISRN Urol. 2011;2011:431951. doi: 10.5402/2011/431951. Epub 2011 Sep 14. PMID 22235380